CLINICAL TRIAL: NCT06672289
Title: Comparison of the Analgesic Effectiveness of Pericapsular Nerve Block and Suprainguinal Fascia Iliac Block Application in Patients Undergoing Hip Arthroscopy
Brief Title: Comparison of the Analgesic Effectiveness of Pericapsular Nerve Block and Suprainguinal Fascia Iliac Block Application
Status: Not yet recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Recep Aksu, Prof. Dr. Recep AKSU, TC Erciyes University
Other Study IDs: 2024/162
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Hip Surgery
Keywords: hip arthroscopy; PENG block; Suprainguinal Fascia Iliaca Block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pericapsular Nerve Block (PENG): Patients will be monitored with routine monitoring under operating room conditions. After the patient's baseline VAS score and vital signs are recorded, patients will be intubated after induction of general anesthesia. After the site is cleaned, pericapsular nerve block (PENG) will be applied under USG guidance. After the procedure, the patient will be transferred to the surgical team for positioning. Blood pressure and pulse values will be recorded after the procedure and at the 30th minute of surgery. After the patients wake up, another anesthesiologist in the recovery unit will rate the pain of patients in both groups on a scale of 0-10, using the Visual Analogue Scale (VAS) to describe their pain intensity. Heart rates and noninvasive blood pressures of patients taken to the recovery unit will be measured and recorded.
- Suprainguinal Fascia Iliaca Block (SFIB): Patients will be monitored with routine monitoring under operating room conditions. After the patient's baseline VAS score and vital signs are recorded, patients will be intubated after induction of general anesthesia. After the site is cleaned, suprainguinal fascia iliaca block (SFIB) will be applied under USG guidance. After the procedure, the patient will be transferred to the surgical team for positioning. Blood pressure and pulse values will be recorded after the procedure and at the 30th minute of surgery. After the patients wake up, another anesthesiologist in the recovery unit will rate the pain of patients in both groups on a scale of 0-10, using the Visual Analogue Scale (VAS) to describe their pain intensity. Heart rates and noninvasive blood pressures of patients taken to the recovery unit will be measured and recorded.

SUMMARY:
Suprainguinal Fascia iliac compartment outlet and Pericapsular nerve reduction, which is a routinely successful method for postoperative analgesia in anesthesia practice; the aim is to investigate information regarding postoperative pain level, analgesic consumption, patient satisfaction and discharge time after arm arthroscopy.

DETAILED DESCRIPTION:
Patients will be monitored with routine monitoring under operating room conditions. After the patient's baseline VAS score and vital signs are recorded, patients will be intubated after induction of general anesthesia. After the site is cleaned, a pericapsular nerve block (PENG) or suprainguinal fascia iliac block (SFIB) will be performed under USG guidance. After the procedure, the patient will be transferred to the surgical team for positioning. Blood pressure and pulse values will be recorded after the procedure and at the 30th minute of surgery.

After the patients wake up, another anesthesiologist in the recovery unit will rate the pain of patients in both groups on a scale of 0-10, using the Visual Analogue Scale (VAS) to describe their pain intensity. Heart rates and noninvasive blood pressures of patients taken to the recovery unit will be measured and recorded. Patient-controlled Analgesia (PCA) will be used for postoperative analgesia for all patients, as is routinely done, and total analgesic consumption will be evaluated. Hemodynamic data, VAS pain scores, and observed hemodynamic data of the patients were examined at 30 minutes, 60 minutes, 90 minutes, 120 minutes, and 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 hours in the postoperative period. Side effects will be recorded. The evaluation of the pain occurring when the hip is immobilized (VASd) and when it is moved (VASh) will be made by the anesthesiologist with VAS.

Patients' 24-hour postoperative satisfaction will be evaluated. Within the scope of the study, patients' gender, age, height, weight, ASA risk scores and operation times will be recorded.

In the statistical evaluation of the study; Analgesic consumption during the procedure, VAS scores, and analgesic consumption and patient satisfaction in the postoperative period will be evaluated and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 and under the age of 65 who will undergo hip arthroscopy
* ASA I-II group patients
* Patients without allergies

  * Patients without psychiatric disorders
* Patients without opioid addiction
* Patients who have the ability to use the patient-controlled analgesia (PCA) device and perform VAS scoring
* Patients with no contraindications for peripheral blocks

Exclusion Criteria:

* Patients who do not want to participate in the study
* Patients with uncontrolled hypertension
* Patients with chronic pain or receiving pain treatment,
* Significant Cardiac Disorder (Coronary Artery Disease, Arrhythmia, Electrocardiography Anomaly, Heart Failure, etc.)
* Patients with Diabetes Mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders will be included this study
Study Population: Patients over the age of 18 and under the age of 65 who will undergo hip arthroscopy
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score | 2-3 hours after surgery
  A Visual Analogue Scale (VAS) is one of the pain rating scales. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. From the patient's perspective, this spectrum appears continuous; their pain does not take discrete jumps, as a categorization of none, mild, moderate and severe would suggest the VAS score for grading of pain consists of a 10 centimetres (cm) line with 10 mm (0.01 cm) to each point of the scale and two end-points representing no pain and worst possible pain, where 0 = no pain, 1-3 = mild, 4-6 = moderate and 7-10 = severe pain

IPD SHARING:
Plan to Share IPD: No